CLINICAL TRIAL: NCT06444815
Title: A Phase 1/1b Study of VET3-TGI Administered Alone and in Combination With Pembrolizumab in Patients With Advanced Solid Tumors
Brief Title: A Study of VET3-TGI in Patients With Solid Tumors
Acronym: STEALTH-001
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: KaliVir Immunotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STEALTH-001
Record Dates: First submitted 2024-05-30; First posted 2024-06-06 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Solid Tumor, Adult; Microsatellite Stable Colorectal Cancer; Head and Neck Squamous Cell Carcinoma; Cervical Cancer; Kidney Cancer; Renal Cell Carcinoma; Melanoma Stage IV; Merkel Cell Carcinoma of Skin; Mesothelioma; Non-small Cell Lung Cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Uterine Cervical Neoplasms; Kidney Neoplasms; Carcinoma, Renal Cell; Melanoma; Mesothelioma; Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group A: VET3-TGI alone intratumoral (Experimental): Dose escalation of VET3-TGI alone administered by direct injection into tumor(s) x 4. Booster injections of VET3-TGI are permitted for up to 2 years.
  Interventions: Drug: VET3-TGI
- Group B: VET3-TGI intratumoral in combination with pembrolizumab (Experimental): VET3-TGI will be given in combination with pembrolizumab at the highest tolerated dose from Group A. Pembrolizumab will be administered via intravenous (IV) infusion for up to 2 years.
  Interventions: Drug: VET3-TGI; Drug: Pembrolizumab
- Group C: VET3-TGI alone intravenous (Experimental): Dose escalation of VET3-TGI alone administered by IV infusion x 6. Booster infusions of VET3-TGI are permitted for up to 2 years.
  Interventions: Drug: VET3-TGI
- Group D: VET3-TGI intravenous in combination with pembrolizumab (Experimental): VET3-TGI will be given in combination with pembrolizumab at the highest tolerated dose from Group C. Pembrolizumab will be administered via intravenous (IV) infusion for up to 2 years.
  Interventions: Drug: VET3-TGI; Drug: Pembrolizumab

INTERVENTIONS:
Drug: VET3-TGI — Oncolytic vaccinia virus engineered with immunomodulatory transgenes
Drug: Pembrolizumab — anti-pd1 antibody
  Arms: Group B: VET3-TGI intratumoral in combination with pembrolizumab; Group D: VET3-TGI intravenous in combination with pembrolizumab

SUMMARY:
VET3-TGI is an oncolytic immunotherapy designed to treat advanced cancers. VET3-TGI has not been given to human patients yet, and the current study is designed to find a safe and effective dose of VET3-TGI when administered by direct injection into tumor(s) (called an intratumoral injection) or when given intravenously (into the vein) both alone and in combination with pembrolizumab in patients with solid tumors (STEALTH-001).

DETAILED DESCRIPTION:
VET3-TGI was changed in a laboratory to infect and kill cancer cells, leaving healthy cells alone. This is a Phase 1 dose escalation (and expansion) study with VET3-TGI administered by direct injection into tumor(s) or by intravenous infusion. The dose escalation has 4 groups: the first group (Group A) will determine the highest tolerated dose of VET3-TGI when injected into tumor(s); the second group (Group C) will determine the highest tolerated dose of VET3-TGI when infused into the vein. The third and fourth groups (Group B and D) will combine VET3-TGI with pembrolizumab. These groups will begin at the highest tolerated dose determined in Group B and Group D, respectively.

Once the highest tolerated dose is found for each of these groups, that dose may be expanded to up to 15 additional patients to better examine the efficacy of VET3-TGI.

ELIGIBILITY:
Key Inclusion Criteria:

* Have pathologically confirmed, advanced, unresectable, or metastatic solid tumors. Preferred indications include, but are not limited to, breast carcinoma, bladder carcinoma, cervical squamous carcinoma, colorectal carcinoma, esophageal carcinoma, head and neck squamous carcinoma, renal cell carcinoma, ovarian carcinoma, sarcoma, thymoma, and uterine carcinoma.
* Failed, intolerant to, or refused potentially curative treatment options, including but not limited to, standard of care molecularly targeted agents, immunotherapy (e.g., anti -pembrolizumab/PDL1 antibodies), and chemotherapy
* Measurable disease as per RECIST 1.1 criteria
* At least one tumor amenable to safe ITu injections and/or biopsies
* ECOG performance status 0 or 1
* Demonstrate adequate organ function
* Must be willing to comply with all protocol procedures and adhere to post-treatment care instructions

Additional Inclusion criteria exist

Key Exclusion Criteria:

* Prior systemic therapy washout (dependent upon the therapy)
* Requires use of anti-platelet or anti-coagulant therapy that cannot be safely suspended for per protocol biopsies or intra-tumoral injections.
* CNS metastases and/or carcinomatous meningitis that have not been completely resected or completely irradiated.
* Prior history of myocarditis
* Known HIV/AIDS, active HBV or HCV infection.
* Receiving high dose immunosuppressive medication or has a significant immunodeficiency (e.g. transplant recipient, etc).

Additional Exclusion criteria exist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events with VET3-TGI alone or in combination with pembrolizumab | 108 months
  Percentage of patients with adverse events by grade as determined by NCI CTCAE v5.0
Incidence of dose limiting toxicities reported with VET3-TGI alone or in combination with pembrolizumab | 4 weeks
  Number of dose limiting toxicities, as defined in the protocol, by dose group
Determine the recommended Phase 2 dose | 4 weeks
  he highest dose of VET3-TGI in each group that can be administered where fewer than 2 patients have a dose-limiting safety event alone or when combined with pembrolizumab as assessed by NCI CTCAE v.5.0 during the Phase 1 dose escalation

SECONDARY OUTCOMES:
Efficacy assessment: overall response rate (ORR) | 108 months
  The number and proportion of patients with a partial response (PR) or complete response (CR) on imaging by RECIST 1.1
Efficacy assessment: Duration of response (DOR) | 108 months
  Median duration of response in patients with a CR or PR
Efficacy assessment: disease control rate (DCR) | 108 months
  The number and proportion of patients with stable disease (SD), or a partial response (PR) or complete response (CR) on imaging by RECIST 1.1
Efficacy assessment: Time to tumor progression (TTP) | 108 months
  Median time until patient disease progression (PD)
Efficacy assessment: Progression free survival (PFS) | 108 months
  Median duration of progression free survival of subjects
Overall survival | 108 months
  median duration of survival across all subjects
Immune changes in tissue and blood | 6 weeks
  number of subject tissue samples with immune cell infiltrates and heat map changes in the molecular signature of tissue samples
VET3-TGI delivery and replication kinetics | 6 weeks
  Number of subject tissues with positive VET3-TGI gene signatures denoting delivery and complete replication of VET3-TGI

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - UC Irvine Health, Orange, California
  - University of Miami, Miami, Florida
  - Community Health Network, Indianapolis, Indiana
  - UPMC- Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Mary Crowley Cancer Research, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
Data is aggregated.